CLINICAL TRIAL: NCT06624085
Title: A Phase Ib Study Evaluating the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of Glofitamab in Combination With Gemcitabine Plus Oxaliplatin in U.S. Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Study Evaluating the Safety and Efficacy of Glofitamab + Gemcitabine + Oxaliplatin in U.S. Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO44900
Record Dates: First submitted 2024-10-01; First posted 2024-10-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — glofitamab; tocilizumab; obinutuzumab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemcitabine + Glofitamab + Oxaliplatin (Experimental): Participants will receive a single dose of intravenous (IV) obinutuzumab pretreatment 7 days prior to the first dose of glofitamab, followed by up to 8 cycles of glofitamab + gemcitabine + oxaliplatin. This will be followed by up to 4 cycles of glofitamab monotherapy, for a total of up to 12 cycles of glofitamab (cycle length = 21 days).
  Interventions: Drug: Glofitamab; Drug: Tocilizumab; Drug: Obinutuzumab; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Glofitamab — Participants will receive IV glofitamab for up to 12 cycles (cycle length = 21 days)
Drug: Tocilizumab — Participants will receive IV tocilizumab as needed to manage cytokine release syndrome (CRS)
Drug: Obinutuzumab — Participants will receive IV obinutuzumab pretreatment
Drug: Gemcitabine — Participants will receive IV gemcitabine for up to 8 cycles (cycle length = 21 days)
Drug: Oxaliplatin — Participants will receive IV oxaliplatin for up to 8 cycles (cycle length = 21 days)

SUMMARY:
The purpose of the study is to evaluate glofitamab + gemcitabine + oxaliplatin in participants in the United States, including under-represented racial and ethnic populations, that have relapsed or refractory (R/R) diffuse large B-cell lymphoma (DLBCL).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed DLBCL, not otherwise specified (NOS)
* Relapsed (disease that has recurred following a response that lasted ≥ 6 months after completion of the last line of therapy) or refractory ( disease that did not respond to or that progressed < 6 months after completion of the last line of therapy) disease
* At least one prior line of systemic therapy
* Participants who have failed only one prior line of therapy must not be a candidate for high-dose chemotherapy followed by autologous stem cell transplant (ASCT)
* At least one bi-dimensionally measurable (> 1.5 cm) nodal lesion, or one bi-dimensionally measurable (> 1 cm) extranodal lesion, as measured on CT scan
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2

Exclusion Criteria:

* Prior enrollment in Study GO41944 (STARGLO; NCT04408638)
* Participant has failed only one prior line of therapy and is a candidate for stem cell transplantation
* History of transformation of indolent disease to DLBCL
* High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements, and high-grade B-cell lymphoma NOS, as defined by 2016 WHO guidelines
* Primary mediastinal B-cell lymphoma
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies (or recombinant antibody-related fusion proteins) or known sensitivity or allergy to murine products
* Prior treatment with glofitamab or other bispecific antibodies targeting both CD20 and CD3
* Prior treatment with gemcitabine or oxaliplatin
* Peripheral neuropathy or paresthesia assessed to be Grade >/= 2 according to NCI CTCAE v5.0 at enrollment
* Treatment with radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy, or any investigational agent for the purposes of treating cancer within 2 weeks prior to first study treatment
* Treatment with monoclonal antibodies for the purposes of treating cancer within 4 weeks prior to first study treatment
* Primary or secondary CNS lymphoma at the time of recruitment or history of CNS lymphoma
* Prior CNS involvement that has been definitively treated and confirmed via MRI or cerebrospinal fluid analysis to be in complete remission is permissible
* Current or history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* History of other primary malignancy, with exceptions defined by the protocol
* Significant or extensive cardiovascular disease, or significant pulmonary disease
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (exclusing fungal infections of nail beds) at study enrollment or any major episode of infection within 4 weeks prior to the first study treatment
* Documented severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 6 months of first study treatment, or positive SARS-CoV-2 test within 7 days prior to enrollment
* Suspected or latent tuberculosis
* Positive test results for hepatitis B (HBV) or hepatitis C (HCV)
* Known or suspected chronic active Epstein-Barr viral infection
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* Known history of progressive multifocal leukoencephalopathy
* Prior solid organ transplantation
* Prior allogenic stem cell transplant
* Active autoimmune disease requiring treatment
* Prior treatment with systemic immunosuppressive medications within 4 weeks prior to first dose of study treatment
* Ongoing systemic corticosteroid use which, in the opinion of the investigator, puts the patient at increased risk of steroid-related iatrogenic adrenal insufficiency
* Recent major surgery (within 4 weeks before the first study treatment) other than for diagnosis
* Clinically significant history of cirrhotic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 3 years
Complete response (CR) rate | Up to 3 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
Duration of response (DOR) | From the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (up to 3 years)
Duration of CR | From the first occurrence of a documented CR to disease progression or death from any cause, whichever occurs first (up to 3 years)
Progression-free survival (PFS) | From enrollment to the first occurrence of disease progression or death from any cause, whichever occurs first (up to 3 years)
Overall Survival (OS) | From enrollment to date of death from any cause (up to 3 years)
Serum concentration of glofitamab | Up to 3 years
Incidence of anti-drug antibodies to glofitamab | Baseline up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- United States (15):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - University of California Los Angeles (UCLA) - Cancer Care - Santa Monica, Santa Monica, California
  - Georgetown University, Washington D.C., District of Columbia
  - AdventHealth Cancer Institute, Orlando, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Illinois Cancer Center, Chicago, Illinois
  - Kansas City VA Medical Center, Kansas City, Kansas
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christus Health - Christus St. Vincent Regional Medical Center, Santa Fe, New Mexico
  - East Carolina University, Greenville, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Renovatio Clinical - El Paso, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas
  - Renovatio Clinical, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No